CLINICAL TRIAL: NCT07179016
Title: A Pragmatic, Randomized Controlled Trial of a Auricular Point Acupressure - Self-Management (APA-SM) Program for Chronic Musculoskeletal Pain Among Rural Populations.
Brief Title: Evaluating the Auricular Point Acupressure-Self Management Program for Chronic Musculoskeletal Pain Among Rural Populations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jennifer Kawi, Distinguished Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-SN-25-0443
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain (Back / Neck); Chronic Pain Management; Chronic Knee Pain; Joint Pain
Keywords: Chronic Pain; Rural population; Self-management; Chronic musculoskeletal pain; Auricular point acupressure
MeSH Terms: conditions — Chronic Pain; Arthralgia | interventions — Glutamyl Aminopeptidase; Self-Management

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remote APA-SM Training (Experimental): APA-SM self-guided with remote training
  Interventions: Behavioral: Auricular Point Acupressure (APA) - Self Management (SM)
- In-person APA-SM Training (Experimental): APA-SM with in-person training
  Interventions: Behavioral: Auricular Point Acupressure (APA) - Self Management (SM)
- Pain Education (Active Comparator): Education Control
  Interventions: Behavioral: Education Control

INTERVENTIONS:
Behavioral: Auricular Point Acupressure (APA) - Self Management (SM) — APA is a noninvasive and needle-free pain management therapy based on the principles of acupuncture. The APA-SM intervention program is aimed to manage chronic musculoskeletal pain leveraging a mobile app containing APA videos and remote vs in-person guidance or coaching to practice APA based on APA study assignment.
  Arms: In-person APA-SM Training; Remote APA-SM Training
Behavioral: Education Control — Education Control group receive an app but the content will be specific to pain and self-management (no APA content) and they practice pain self-management skills (no APA practice).
  Arms: Pain Education

SUMMARY:
The investigators will test an Auricular Point Acupressure Self-Management (APA-SM) program integrated into rural primary and specialty care and rural communities for chronic musculoskeletal pain (CMP). To maximize self-management of pain, the investigators developed a smartphone app which will allow the participants to learn to self-administer APA. The investigators will have 3 arms (APA-SM self-guided with remote training, APA-SM with in-person training, and Education Control) with 231 participants per arm (total=693 for 3 arms). The investigators will evaluate the clinical effectiveness of our 4-week APA-SM intervention compared to control in primary outcomes (pain intensity, pain interference, activity), secondary outcomes (HEAL Clinical Pain Core common data elements), and analgesic use up to 6 months follow-up.

DETAILED DESCRIPTION:
The investigators integrated ecological momentary assessment into our app to measure real-world outcomes resulting in participants being able to self-monitor their progress, using this as an innovative behavior change strategy based on Bandura's self-efficacy, successfully initiating and maintaining behavior change. The primary endpoint will be immediate post-intervention with secondary endpoints at 1-month, 3-month, and 6-month follow-ups after the intervention. The investigators will also evaluate implementation outcomes and cost-effectiveness. Our long-term goal is to increase the access and scalability of evidence-based interventions while addressing pain care disparities for rural individuals with limited resources and/or endure long distances to specialty pain care. Study recruitment will be 3 1/2 to 4 years followed by data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Receive any pain management for CMP (neck, back, shoulder, hands, hips, knees, feet)
* Have CMP ≥ 4 on a scale of 0-10 that has persisted for at least 3 months or has resulted in pain on at least half the days in the past 6 months

Exclusion Criteria:

* Severe ear skin disorder (Diagnosed with conditions e.g., eczema, lupus with skin involvement) which often require medical intervention and severe allergy to tape
* Inability or unwillingness to provide informed consent
* Use of some type of hearing aid where size may obstruct seed placement
* Not living in rural area

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 693 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain as assessed by the pain, enjoyment of life, general activity (PEG) survey | Baseline, post intervention (4 weeks after baseline), 1 month, 3 months, 6 months
  This is a three-item questionnaire and each is scored from 0 (no pain) to 10(worst pain) for a maximum score of 30. Higher score indicating worse outcome

SECONDARY OUTCOMES:
Change in pain as assessed by the Pain Catastrophizing Scale (PCS6) | Baseline, post intervention (4 weeks after baseline)
  This is a six-item questionnaire and each is scored from 0 (not at all) to 4 (all the time) for a maximum score of 24. Higher score indicating greater pain catastrophizing.
Change in fear-avoidance beliefs as assessed by the Fear-Avoidance Beliefs Questionnaire (FABQ) | Baseline, post intervention (4 weeks after baseline)
  This is a 16-item questionnaire. Each item is scored from 0 (completely disagree) to 6 (completely agree) for a maximum score of 96. Higher score indicating greater fear-avoidance beliefs.
Change in depression as assessed by the Patient Health Questionnaire (PHQ2 ) | Baseline, post intervention (4 weeks after baseline)
  This is a two-item questionnaire and each is scored from 0 (not at all) to 3(nearly every day) for a maximum score of 6. Higher score indicating greater depression.
Change in anxiety as assessed by the Generalized Anxiety Disorder (GAD2) | Baseline, post intervention (4 weeks after baseline)
  This is a two-item questionnaire and each is scored from 0 (not at all) to 3 (nearly every day) for a maximum score of 6. Higher score indicating more anxiety.
Change in severity of pain and its impact on functioning as assessed by the Brief Pain Inventory (BPI) Short From | Baseline, post intervention (4 weeks after baseline)
  This consist of six-item questionnaire regarding pain severity and nine-item questionnaire regarding pain interference. Higher score indicates greater pain severity and interference.
Change in physical function as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function short form 6b (SF6b) | Baseline, post intervention (4 weeks after baseline)
  This is a six-item questionnaire and each is scored from 1 (unable to do) to 5 (without any difficulty) for a maximum score of 30. Higher score indicates better physical function.
Change in disability as assessed by the Roland Morris Disability Questionnaire (RMDQ) | Baseline, post intervention (4 weeks after baseline)
  This is a 24-item questionnaire and each is scored 0 (no) or 1 (yes) for a maximum score of 24. Higher score indicates greater disability.
Change in sleep duration as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) for Sleep 6a (+Sleep Duration) | Baseline, post intervention (4 weeks after baseline)
  This is a six-item questionnaire and each is scored from 1 (very good) to 5 (very poor) for a maximum score of 30. Higher scores indicate worse sleep disturbance. It also includes an additional single item (+Sleep Duration) assessing hours and minutes of sleep per night. Higher values indicates longer sleep duration.
Change in pain self-efficacy influenced by pain as assessed by the Pain Self-Efficacy Questionnaire 2 item Short Form (PSEQ2) | Baseline, post intervention (4 weeks after baseline)
  This is a two-item questionnaire and each is scored from 0 (not at all confident) to 6 (completely confident) for a maximum score of 12. Higher score indicating greater pain self-efficacy.
Change in substance use as assessed by the Tobacco, Alcohol, Prescription medication, and other Substance (TAPS1) Substance Use Screener | Baseline, post intervention (4 weeks after baseline)
  This is a five-item questionnaire and each is scored from 0 (daily or almost daily) to 4 (never) for a maximum score of 20. Higher score indicates lower substance use.
Change in quality of life as assessed by the World Health Organization Quality of Life 2 item (WHOQOL-2) | Baseline, post intervention(4 weeks after baseline)
  This is a two-item questionnaire and each is scored from 1 (very poor/dissatisfied) to 5 (very good/satisfied) for a maximum score of 10. Higher score indicating better quality of life.
Change in positive outlook as assessed by the Healing Encounters and Attitudes Lists (HEAL) | Baseline, post intervention(4 weeks after baseline)
  This is a six-item questionnaire and each is scored from 1 (not at all) to 5 (very much) for a maximum score of 30. Higher score indicates greater positive outlook.
Change in treatment expectancy as assessed by the Healing Encounters and Attitudes Lists (HEAL) | Baseline, post intervention(4 weeks after baseline)
  This is a six-item questionnaire and each is scored from 1 (not at all) to 5 (very much) for a maximum score of 30. Higher score indicates greater treatment expectancy.
Change in attitude towards complement alternative medicine (CAM) as assessed by the Healing Encounters and Attitudes Lists (HEAL) | Baseline, post intervention (4 weeks after baseline)
  This is a six-item questionnaire and each is scored from 1 (not at all) to 5 (very much) for a maximum score of 30. Higher score indicates more positive attitude toward CAM.
Change in analgesics and opioid use as assessed by the Ecological Momentary Assessment (EMA) diary | Baseline, post intervention (4 weeks after baseline)
  Daily self-reported analgesic and opioid use (type, dose, frequency) recorded via EMA diary

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kawi, PhD, MSN, FNP-BC, CNE, FAAN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (3):
- United States (3):
  - University of South Carolina, Columbia, South Carolina
  - University of North Texas Health Science Center at Fort Worth, Fort Worth, Texas
  - The University of Texas Health science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
We have a Data Management and Sharing Plan and will comply with the policy set forth by NIH.